CLINICAL TRIAL: NCT01203904
Title: Pulmicort Turbuhaler 100/200 Specific Clinical Experience Investigation for Long Term Use in Pediatrics
Brief Title: Pulmicort Turbuhaler 100/200 Specific Clinical Experience Investigation
Acronym: PEACE-Peds
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D525AL00001
Record Dates: First submitted 2010-09-06; First posted 2010-09-17 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma, Pulmicort, long term use, pediatrics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pulmicort

SUMMARY:
The purpose of this study is to confirm the safety profile for long term treatment in children aged 5 years and <15 years on bronchial asthma in daily clinical usage/Effect on growth rate. Effect on adrenal function. Development of infection diseases by diseases type.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Pulmicort Turbuhaler for the first time due to bronchial asthma and children of >= 5 years and < 15 years old age at the start of study treatment

Exclusion Criteria: -None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Pulmicort Turbuhaler for the firtst time due to bronchial asthma and children of >= 5 years and < 15 years old age at the start of study treatment
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence. We will investigate, intensively, development of Adverse Drug Reactions, especially infections. Detection of Adverse Drug Reactions unexpected from the Precautions for use. | Two years
Effects on growth rate and the adrenal cortical function, development of infections | Two years

SECONDARY OUTCOMES:
Variation of the asthma control status (total of JPAC：Japanese Pediatric Asthma Control Program score) from the baseline score. | Two years
Variation of the parental questionnaire (score by factor) from the baseline score. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, Study Director — AstraZenecaKK
Locations (37):
- Japan (37):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Nagano
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Yamagata
  - Research Site, Yamaguchi

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=499&filename=Pulmicort-sCEI_synopsis_20160606.pdf